CLINICAL TRIAL: NCT01689480
Title: Prospective Study for 24-months of Physical Training Introduced in Lifestyle of Patients With Facioscapulohumeral Dystrophy : Tolerance, Sustainability and Efficiency of Unsupervised Training Program.
Brief Title: Prospective Study for 24-months of Physical Training Introduced in Lifestyle of Patients With FSHD : Tolerance, Sustainability and Efficiency of Unsupervised Training Program.
Acronym: FSHD2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 1108153; 2011-A01186-35 (Other: AFSSAPS)
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Muscular Dystrophy, Facioscapulohumeral
Keywords: Muscular Dystrophy; Facioscapulohumeral; Physical training; Exercise
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FSHD training: Only the patients who have participated to the FSHD1 study (NCT01116570) can be included in this study.
  Interventions: Other: FSHD training

INTERVENTIONS:
Other: FSHD training — The training will consist in 3 sessions of 35 min of training per week at home on an ergocycle. The training will be divided in (i) 2 sessions of 30 min aerobic exercises at a constant but moderate (60% of maximal aerobic power, MAP) intensity followed with 5 sets of 10 revolutions at near-maximal intensity and (ii) an interval-training session. This latter session will consist in 5 min warm-up at 40% MAP followed by 5 times 1 min at 80% MAP (recovery = 4 min at 40% MAP) followed by 5 min of active recovery. A systematic supervision of the sessions by the coach will be performed by phone, by using the heart rate recordings and values of Analogic Visual Scale for pain and fatigue.

SUMMARY:
It is now accepted that physical activity is not deleterious in myopathies, including muscular dystrophies. In patients suffering from facioscapulohumeral dystrophy (FSHD), aerobic training has been reported to be associated with physiological and functional positive effects without alteration in quality of life. Van der Kooi et al. (2005) and Cup et al. (2007) studies suggest that the combination of endurance and strength trainings is even more relevant. However, only a few controlled and randomized studies have been conducted on this topic and the impact of such training programs on skeletal muscle regenerative capacities has not been addressed yet. Moreover, due to the fact that training programs are mainly performed on short-term supervised periods, there is a lack of knowledge regarding long-term effects, patient's autonomy and whether or not practice of regular exercise can be maintained in patient's daily life. Also, only a few experiments report an integrative view of potential benefits of such programs on functional, biological and quality of life.

DETAILED DESCRIPTION:
The present project is the second phase of a study for which the first phase currently financed by AFM is in progress and aims to establish a program of adapted physical training performed at the patient's home under supervision. This program was developed in order to try to meet the two following requirements: 1) to be compatible with the daily professional/social activity of patients so it can be integrated in their life routine; 2) to be intense enough so functional benefits can be induced. The first phase is a controlled and randomized study where patients with FSHD participate in a 6-months supervised training program combining aerobic and strength training sessions on an ergocycle.

This second phase of our research project aims to evaluate whether a long-term integration of this adapted training program into patients' lifestyle is possible. The same tools, same method and same measurements of training program will be used with remote monitoring, less frequent as it was in the first phase, over a period of 24 months. This second experimental work will also be based on multi-factorial evaluations, i.e. biological, physiological, functional, and quality of life questionnaires and remains collaboration between Universities of Saint Etienne (L. Féasson), Grenoble (B Wuyam) and Örebro (F Kadi) within the Rhône-Alpes Reference Centre for Rare Neuromuscular Diseases (JC Antoine).

ELIGIBILITY:
Inclusion Criteria:

* Included in the FSHD1 study
* Social Security regimen affiliated
* Consent form signed

Exclusion Criteria:

* Severe cardiac or respiratory insufficiency
* Cardiac pacemaker
* Morbid obesity (BMI upper to 35)
* Anti platelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with facioscapulohumeral dystrophy and who have participated to the FSHD1 study
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
patient's compliance | at 24 months
  Number of adapted physical activity sessions conducted over 2 years in patients with FSHD based on a theoretical program of three weekly sessions. A session will be considered valid based on the collection 1) time physical activity actually performed and 2) its intensity, both recorded from the cycle ergometer and a heart rate record.

CONTACTS AND LOCATIONS:
Overall Officials: Léonard FEASSON, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (2):
- France (2):
  - CHU de Grenbole, Grenoble
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No